CLINICAL TRIAL: NCT01688310
Title: A Randomized Controlled Trial of Open Surgical vs. Minimally-invasive Voluntary Adult Male Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Católica de Moçambique (Other)
Collaborators: University of Pittsburgh (Other); Catholic University of Mozambique (Other)
Responsible Party: Principal Investigator, Dr. Peter Millard, Clinical Director of the Health Center, Universidade Católica de Moçambique
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO11080657
Record Dates: First submitted 2012-08-27; First posted 2012-09-19 (Estimated); Results first posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-06

CONDITIONS: Surgical Technique
Keywords: Gomco clamp instrument; Tissue adhesive; Open surgical circumcision; Minimally-invasive circumcision
MeSH Terms: interventions — Tissue Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open surgical circumcision (Active Comparator): Open surgical techniques, which are commonly used for circumcision in Mozambique, require good surgical skills and minor complications are common.
  Interventions: Procedure: Open surgical circumcision
- Gomco clamp with tissue adhesive (Experimental): Coupling removal of the foreskin with the Gomco clamp followed by wound sealing with tissue adhesive results in a procedure that can be performed by generalist doctors using the same technique in all age groups.
  Interventions: Procedure: Gomco Clamp with Tissue Adhesive

INTERVENTIONS:
Procedure: Gomco Clamp with Tissue Adhesive — According to WHO (2011), the Gomco clamp has "…an impeccable safety record. In the USA, where it is estimated that well over 1 million neonates are circumcised each year, the Gomco clamp has become the leading instrument used to perform non-ritual male circumcision." Tissue adhesive is widely used in multiple areas of medicine; specifically, multiple observational studies and RCTs have shown cyanoacrylate tissue adhesives to be superior to suture closure in VMMC.
  Arms: Gomco clamp with tissue adhesive
Procedure: Open surgical circumcision — The World Health Organization, in its Manual for Male Circumcision under Local Anaesthesia, describes three open surgical techniques (forceps assisted, dorsal slit and sleeve technique), all three of which involve (a) exposure of subcutaneous tissues and (b) suturing for hemostasis and for skin closure.
  Arms: Open surgical circumcision

SUMMARY:
This proposed randomized controlled trial will provide important data which will inform and enable the Mozambican government and global health programs to more effectively scale-up circumcision services. The investigators postulate that voluntary medical male circumcision using the Gomco clamp coupled with tissue adhesive meets WHO criteria for the ideal method: it is much easier to learn, faster, safer for both surgeons and patients, heals sooner, and is more cost effective than any other currently available technique.

DETAILED DESCRIPTION:
Voluntary medical male circumcision (VMMC) is a priority preventive intervention and Mozambique is a priority country for VMMC scale-up. PEPFAR recently estimated that one HIV infection would be prevented between now and 2025 for every seven circumcisions performed in Mozambique. Sofala Province, where the study will be conducted, has an HIV prevalence of 13% among men and 18% among women. Approximately 8% of men aged 15-49 in Sofala Province, where the study will take place, are currently circumcised.

In spite of their widely acknowledged drawbacks, open surgical techniques are the only VMMC techniques the President's Emergency Plan for AIDS Relief (PEPFAR) program currently allows in Africa. According to the Framework for Clinical Evaluation of Devices for Adult Male Circumcision (WHO, 2011): "WHO and other health authorities wish to identify one or more devices that (a) would make the VMMC safer, easier, and quicker; (b) would have more rapid healing than current methods and/or might entail less risk of HIV transmission in the post-operative period; (c) could be performed safely by health-care providers with a minimal level of training; and (d) would be cost-effective compared to standard surgical methods for male circumcision scale up."

This proposed randomized controlled trial will provide important data which will inform and enable the Mozambican government and PEPFAR to more effectively scale-up circumcision services. The investigators postulate that VMMC using the Gomco clamp coupled with tissue adhesive meets WHO criteria for the ideal method: it is much easier to learn, faster, safer for both surgeons and patients, heals sooner, and is more cost effective than any other currently available technique.

The investigators propose a randomized controlled trial (RCT) comparing this minimally-invasive circumcision technique to the open surgical technique:

* Gomco clamp with tissue adhesive: 100 men
* Open surgical circumcision: 100 men

The Gomco clamp is an FDA-approved device widely used in the US, but there are few data on its use in Africa. Tissue adhesive is widely used in multiple areas of medicine; specifically, multiple observational studies and RCTs have shown cyanoacrylate tissue adhesives to be superior to suture closure in circumcision in boys. The investigators refer to Gomco clamp circumcision coupled with tissue adhesive as a 'new' technique because these two independently-validated components have only been coupled in observational studies among men, and in randomized controlled trials among pre-pubertal boys, but never before in an RCT among adult men. The open surgical method is PEPFAR-approved and will serve as the control intervention.

Population: Men > 18 years of age who desire male circumcision Sample size: 200 (100 men in each group) Study design: Randomized controlled trial Intervention: Gomco clamp circumcision plus tissue adhesive vs. open surgical circumcision Follow-up visits: 2 days, 7 days, 14 days and 28 days. Optional 42 day follow-up if not completely healed by 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men > 18 years of age requesting circumcision
* No penile anatomical abnormalities or infections
* Able to provide informed consent to participate
* Willing to participate in follow-up visits

Exclusion Criteria:

* Current illness
* Penile abnormality or infection which contraindicates or would complicate circumcision
* History of bleeding disorder
* Past reaction to local anesthetic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Millard, MD, PhD, Principal Investigator — Universidade Catholic de Mozambique
Locations (1):
- Centro de Saúde São Lucas, UCM, Beira, Sofala, Mozambique

REFERENCES:
- [Background] Gray RH, Kigozi G, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chaudhary MA, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Williams CF, Opendi P, Reynolds SJ, Laeyendecker O, Quinn TC, Wawer MJ. Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial. Lancet. 2007 Feb 24;369(9562):657-66. doi: 10.1016/S0140-6736(07)60313-4. PMID 17321311
- [Background] Bailey RC, Muga R, Poulussen R, Abicht H. The acceptability of male circumcision to reduce HIV infections in Nyanza Province, Kenya. AIDS Care. 2002 Feb;14(1):27-40. doi: 10.1080/09540120220097919. PMID 11798403
- [Background] Lagarde E, Dirk T, Puren A, Reathe RT, Bertran A. Acceptability of male circumcision as a tool for preventing HIV infection in a highly infected community in South Africa. AIDS. 2003 Jan 3;17(1):89-95. doi: 10.1097/00002030-200301030-00012. PMID 12478073
- [Background] Scott BE, Weiss HA, Viljoen JI. The acceptability of male circumcision as an HIV intervention among a rural Zulu population, Kwazulu-Natal, South Africa. AIDS Care. 2005 Apr;17(3):304-13. doi: 10.1080/09540120412331299744. PMID 15832878
- [Background] Mattson CL, Bailey RC, Muga R, Poulussen R, Onyango T. Acceptability of male circumcision and predictors of circumcision preference among men and women in Nyanza Province, Kenya. AIDS Care. 2005 Feb;17(2):182-94. doi: 10.1080/09540120512331325671. PMID 15763713
- [Background] Halperin DT, Fritz K, McFarland W, Woelk G. Acceptability of adult male circumcision for sexually transmitted disease and HIV prevention in Zimbabwe. Sex Transm Dis. 2005 Apr;32(4):238-9. doi: 10.1097/01.olq.0000149782.47456.5b. No abstract available. PMID 15788922
- [Background] Bailey RC, Egesah O, Rosenberg S. Male circumcision for HIV prevention: a prospective study of complications in clinical and traditional settings in Bungoma, Kenya. Bull World Health Organ. 2008 Sep;86(9):669-77. doi: 10.2471/blt.08.051482. PMID 18797642
- [Background] Kim HH, Goldstein M. High complication rates challenge the implementation of male circumcision for HIV prevention in Africa. Nat Clin Pract Urol. 2009 Feb;6(2):64-5. doi: 10.1038/ncpuro1279. Epub 2008 Dec 23. PMID 19107114
- [Background] Lane V, Vajda P, Subramaniam R. Paediatric sutureless circumcision: a systematic literature review. Pediatr Surg Int. 2010 Feb;26(2):141-4. doi: 10.1007/s00383-009-2475-y. Epub 2009 Aug 26. PMID 19707772
- [Background] Elmore JM, Smith EA, Kirsch AJ. Sutureless circumcision using 2-octyl cyanoacrylate (Dermabond): appraisal after 18-month experience. Urology. 2007 Oct;70(4):803-6. doi: 10.1016/j.urology.2007.07.002. PMID 17991565
- [Background] Kaye JD, Kalisvaart JF, Cuda SP, Elmore JM, Cerwinka WH, Kirsch AJ. Sutureless and scalpel-free circumcision--more rapid, less expensive and better? J Urol. 2010 Oct;184(4 Suppl):1758-62. doi: 10.1016/j.juro.2010.03.081. Epub 2010 Aug 21. PMID 20728122
- [Background] World Health Organization. Male circumcision: Global trends and determinants of prevalence, safety and acceptability, 2007
- [Background] World Health Organization. Manual for Male Circumcision under Local Anaesthesia. 2009.
- [Background] World Health Organization. Manual for early infant male circumcision under local anaesthesia. 2010.
- [Background] World Health Organization. Framework for Clinical Evaluation of Devices for Adult Male Circumcision. 2011.
- [Background] PEPFAR Next Generation Indicators Reference Guide, Vers 1.1, 2009 At www.pepfar.gov/documents/organization/81097.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between October 30, 2012 and February 2, 2013. University teaching clinic.
Pre-assignment Details: 241 interviewed, Excluded (n=41)
  * Inclusion criteria not met (n=19)
    * Under 18 years of age (n=17)
    * Phimosis (n=2)
  * Declined to participate (n=22) 200 were randomized and underwent circumcision in the arm allocated
Groups:
- Open Surgical Circumcision: Open surgical techniques, which are commonly used for circumcision in Subsaharan Africa (and the only technique permitted by PEPFAR), require good surgical skills and minor complications are common.
Period: Overall Study
Arm/Group | Open Surgical Circumcision | Gomco Clamp With Tissue Adhesive
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Surgical Circumcision | Gomco Clamp With Tissue Adhesive | Total
Number analyzed (Participants) | 100 | 100 | 200
Age Continuous [Mean (Standard Deviation); unit: years] | 22.8 (4.9) | 22.3 (4.7) | 22.5 (4.8)
Age, Customized [Number; unit: participants]
  18-20 yrs | 43 | 49 | 92
  21-24 yrs | 26 | 27 | 53
  >=25 yrs | 31 | 24 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 100 | 100 | 200
Region of Enrollment [Number; unit: participants]
  Mozambique | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Duration
Description: Time it takes for procedure from first manipulation of tissue under local anesthesia to dressing.
Time Frame: 1 year
Population: All participants
Measure: Mean (Standard Deviation); unit: Min
Arm/Group | Open Surgical Circumcision | Gomco Clamp With Tissue Adhesive
Number analyzed (Participants) | 100 | 100
Min | 22.5 (6.6) | 12.8 (2.7)

2. Secondary Outcome: Difficulty in Learning and Performing Technique
Description: Evaluated by doctor survey, 5 point Likert scale:
  1. Gomco technique is much easier
  2. Gomco technique is easier
  3. Neutral
  4. Open surgical technique is easier
  5. Open surgical technique is much easier
Time Frame: 1 year
Measure: Median (Full Range); unit: units on Likert scale
Groups:
- Senior Physicians: Physicians who had extensive prior experience performing open surgical circumcisions.
- Junior Physicians: Physicians who had very limited prior experience performing open surgical circumcisions.
Arm/Group | Senior Physicians | Junior Physicians
Number analyzed (Participants) | 4 | 9
units on Likert scale | 2.5 [1 to 5] | 2 [1 to 5]

3. Secondary Outcome: Time Required for Healing
Description: Time required for healing
Time Frame: Within 6 weeks after surgery
Measure: Number; unit: percentage of participants
Arm/Group | Open Surgical Circumcision | Gomco Clamp With Tissue Adhesive
Number analyzed (Participants) | 97 | 96
percentage of participants
  Healed at 2 weeks | 2.1 | 9.4
  Healed at 4 weeks | 87.8 | 87.4
  Healed at 6 weeks | 98.9 | 100

4. Secondary Outcome: Direct Costs
Description: the cost of labor, supplies and equipment
Time Frame: Within 6 weeks after surgery
Reporting Status: Not Posted

5. Secondary Outcome: Pain Experienced
Description: Pain experienced during and after the procedure using Pain Questionnaire with 10 point pain scale (0 signifies no pain and 10 signifies maximal pain)
Time Frame: 2 days after surgery
Measure: Mean (Standard Deviation); unit: units on 10 point pain scale
Arm/Group | Open Surgical Circumcision | Gomco Clamp With Tissue Adhesive
Number analyzed (Participants) | 100 | 100
units on 10 point pain scale | 2.5 (1.9) | 1.8 (1.6)

6. Secondary Outcome: Overall Patient Satisfaction
Description: Patient satisfaction evaluated with patient satisfaction questionnaire using five point Likert scale.
Time Frame: Within 6 weeks after surgery
Measure: Number; unit: participants
Arm/Group | Open Surgical Circumcision | Gomco Clamp With Tissue Adhesive
Number analyzed (Participants) | 99 | 95
participants
  Very satisfied | 70 | 56
  Satisfied | 29 | 39
  Not satisfied | 0 | 0

7. Secondary Outcome: Cosmetic Result
Description: Cosmetic result evaluated by classification of scar line as regular (straight without any irregularity), irregular (not completely straight), or scalloped (with a wavy appearance).
Time Frame: Within 6 weeks after surgery
Measure: Number; unit: participants
Arm/Group | Open Surgical Circumcision | Gomco Clamp With Tissue Adhesive
Number analyzed (Participants) | 93 | 94
participants
  Regular | 54 | 93
  Irregular | 35 | 1
  Scalloped | 4 | 0

8. Other Pre Specified Outcome: Adverse Events
Description: Intraoperative and post-operative adverse events, such as bleeding, hematoma, and infection
Time Frame: 1 yr
Measure: Number; unit: participants
Arm/Group | Open Surgical Circumcision | Gomco Clamp With Tissue Adhesive
Number analyzed (Participants) | 100 | 100
participants
  Mild bleeding | 0 | 4
  Moderate bleeding (suturing required) | 1 | 6
  Hematoma | 3 | 1
  Infection (antibiotic required) | 3 | 7

ADVERSE EVENTS:
Arm/Group | Open Surgical Circumcision | Gomco Clamp With Tissue Adhesive
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 7/100 | 18/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Surgical Circumcision (N=100) | Gomco Clamp With Tissue Adhesive (N=100)
Serious post-operative complication (Surgical and medical procedures) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Surgical Circumcision (N=100) | Gomco Clamp With Tissue Adhesive (N=100)
Mild post-operative bleeding (Surgical and medical procedures) | 0 (0) | 4 (4)
Moderate post-operative bleeding (Surgical and medical procedures) | 1 (1) | 6 (6) — Required suturing to stop bleeding
Hematoma (Surgical and medical procedures) | 3 (3) | 1 (1)
Post-operative infection (Surgical and medical procedures) | 3 (3) | 7 (7) — Required antibiotic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No